CLINICAL TRIAL: NCT04740216
Title: A Randomized Feasibility Trial to Test Exercise Therapy Plus Jaw Device to Prevent Trismus in Patients With Head and Neck Cancer Receiving Radiation-Based Therapy
Brief Title: Effects of Exercise Therapy Adjuvant Device on Head and Neck Cancer Patients in the Treatment of Cancer Therapy Induced Trismus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tsai-Wei Huang, Principal Investigator, Clinical Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B202005159
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Maximum Interincisal Opening
Keywords: trismus; head and neck cancer; radiotherapy; maximum interincisal opening
MeSH Terms: conditions — Trismus; Head and Neck Neoplasms | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise therapy plus jaw device (Experimental): exercise therapy plus jaw device
  Interventions: Behavioral: exercise therapy plus jaw device
- exercise therapy (Placebo Comparator): exercise therapy
  Interventions: Behavioral: exercise therapy

INTERVENTIONS:
Behavioral: exercise therapy plus jaw device — The mouth-opening rehabilitation exercise lasts for twelve weeks, five days a week, three times a day. Subjects can arrange to perform before or after meals according to personal eating time and preferences. The experimental group performs 30 minutes each time, including 20 minutes of stretching exercises. Ten-minute mouth expander assisted passive exercise.
  Arms: exercise therapy plus jaw device
Behavioral: exercise therapy — the control group performed 20-minute stretching exercises each time.
  Arms: exercise therapy

SUMMARY:
Trismus is traditionally considered being a late effect of cancer therapy with functional deficits becoming clear in the first year after completing radiation therapy. These deficits can rapidly progress to a state of functional impairment. The most common treatment for trismus is physical therapy comprising an active range of motion (ROM) exercises, hold and relax techniques. Once trismus has developed, it may be hard to reverse. Thus, prevention with a program of self-care is important for managing this side effect. This study want to test the effect with adjunctive devices plus exercise to prevent trismus.

ELIGIBILITY:
Inclusion Criteria:

1. Age is greater than or equal to 20 years old.
2. Those who are able to communicate in Mandarin and Taiwanese and have no reading or listening or writing disabilities can fill out the questionnaire by themselves or with the assistance of the researcher.
3. Diagnosed with head and neck cancer, and is expected to receive head and neck radiation therapy for the first time.
4. A clear consciousness, no severe cognitive impairment or mental symptoms.
5. Willing to participate in this research and obtain consent.

Exclusion Criteria:

1. People with known temporomandibular joint disorders.
2. The maximum opening degree is less than or equal to 25 mm.
3. Those who have received radiotherapy for the head and neck in the past.
4. Those who have been diagnosed by a physician for poor wound healing after surgery and unable to perform mouth-opening rehabilitation exercises.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-02-10 (Estimated); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The change of maximum interincisal opening (MIO) | baseline, 2 weeks, 4 weeks, 6 weeks, 8weeks, 10 weeks, 12 weeks, 6 months.
  Using Gothenburg Trismus Questionnaire, GTQ to measure the trismus condition and mouth opening

SECONDARY OUTCOMES:
The change of fatigue level | baseline, 2 weeks, 4 weeks, 6 weeks, 8weeks, 10 weeks, 12 weeks, 6 months.
  using the Brief Fatigue Inventory, BFI to measure fatigue level
Quality of life (QOL) | baseline, 2 weeks, 4 weeks, 6 weeks, 8weeks, 10 weeks, 12 weeks, 6 months.
  using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 Head and Neck 35-questions, EORTC-QLQ-C30-H&N35 to meaure QOL